CLINICAL TRIAL: NCT05007379
Title: Cohort Study to Determine the Antitumor Activity of New CAR-macrophages in Breast Cancer Patients' Derived Organoids (CARMA)
Brief Title: Cohort Study to Determine the Antitumor Activity of New CAR-macrophages in Breast Cancer Patients' Derived Organoids
Acronym: CARMA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CARMA-2101
Record Dates: First submitted 2021-08-11; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cell-based immune therapy using modified macrophages is a promising therapeutic approach in breast cancer. The objective of this cohort study is to collect tumor samples to develop patients' derived organoids to test the antitumor activity of newly developed CAR-macrophages. Other biological samples will be collected such as blood to analyze the host inflammatory status.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or more
* Histologically confirmed breast cancer at any stage
* Requiring surgery or tumor biopsy as standard of care
* Any or no systemic treatment
* Signed informaed consent
* Health insurance coverage

Exclusion Criteria:

* Opposed to biospecimen collection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a cohort study conducted in breast cancer patients requiring a surgery or a tumor biopsy as part of their care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Antitumor activity of the CAR-macrophages against organoids from HER2 negative, HER2 low and HER2 positive breast cancers | 24 months
Antitumor activity of the CAR-macrophages compared to non-modified macrophages | 24 months

SECONDARY OUTCOMES:
Antitumor activity of the CAR-macrophages against organoids from early and advanced breast cancers patients | 24 months

IPD SHARING:
Plan to Share IPD: Undecided